CLINICAL TRIAL: NCT04371848
Title: Impact of the COVID-19 Pandemic on Diet Quality and Food Insecurity Among Adults From the Province of Québec in Canada: a NutriQuébec Sub-study
Brief Title: Impact of the COVID-19 Pandemic on Diet Quality and Food Insecurity: a NutriQuébec Sub-study
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-042Phase IIA6/09-04-2020
Record Dates: First submitted 2020-04-22; First posted 2020-05-01 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Eating Habits
Keywords: Eating habits; Web-based prospective cohort study; Lifestyle habits; Diet quality; COVID-19; Food insecurity; Health
MeSH Terms: conditions — Feeding Behavior; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The unprecedented confinement and social distancing rules imposed by the fight against COVID-19 has forced the majority of the population worldwide to stay home for periods of time ranging from weeks to months. Eating habits are undoubtedly perturbed during this period, with consequential impact on food security. Therefore, the primary aim of this NutriQuébec sub-study is to document the impacts of the COVID-19 pandemic on diet quality and food insecurity of adults in the province of Québec in Canada.

NutriQuébec is a web-based prospective cohort study launched in June 2019 whose primary aim is to provide data for the evaluation of the Government Health Prevention Policy on the Québec population's eating habits over the years (NCT04140071). Participants of NutriQuébec are invited to complete on a web-based platform nine core questionnaires on a yearly basis. Questionnaires assess several dimensions related to lifestyle, including eating habits and physical activity habits, as well as a large number of personal characteristics and global health status.

For the purpose of this sub-study, NutriQuebec will invite the 2465 active participants who completed the first-year questionnaires prior to the COVID-19 pandemic to fill out again those questionnaires during the peak period of the confinement period in April and May, 2020. This NutriQuébec sub-study will provide invaluable data on how the COVID-19 pandemic impacts diet quality and food insecurity of adults in the province of Québec.

DETAILED DESCRIPTION:
The 2465 active participants of NutriQuébec who completed the first-year questionnaires prior to the COVID-19 pandemic will be invited to provide informed consent to participate in this sub-study. Once having consented, participants will be invited to complete the core questionnaires by logging into their personal and secured account. Participants will have a three-week period to complete the questionnaires, from April 16 to May 7, 2020.

Core questionnaires in NutriQuébec assess lifestyle habits including eating habits, physical activity habits, sleep quality, tobacco, alcohol and drug habits as well as pandemic behaviors, personal characteristics, food insecurity, health status and health-related quality of life. Most of these questionnaires are based on a one-month recall timeframe, with the exception of the eating habits questionnaires, which is in the form of repeated 24-h recall. For the purpose of this NutriQuébec substudy, questionnaires were adapted to focus on habits during the last 7 days of questionnaire completion, to reflect more specifically the confinement period.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over with a residential address in Québec (Canada)
* Be able to read and understand French or English
* Have access to Internet (with a computer, electronic tablet or cell phone)
* Have an active email address

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in the province of Québec (Canada)
Sampling Method: Non-Probability Sample
Enrollment: 2465 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-05-07 (Actual)

PRIMARY OUTCOMES:
Change in diet quality | 0 to 11 months
  Diet quality during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in food insecurity | 0 to 11 months
  Food insecurity during the study period will be assessed using the series of questions of the Household Food Security Survey Module from the Canadian Community Health Survey (CCHS)-2017

SECONDARY OUTCOMES:
Change in intake of sodium | 0 to 11 months
  Intake of sodium during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in intake of sugar | 0 to 11 months
  Intake of sugar during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in intake of saturated fat | 0 to 11 months
  Intake of saturated fat during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in intake of vegetables and fruits | 0 to 11 months
  Intake of vegetables and fruits during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in intake of dairy products | 0 to 11 months
  Intake of dairy products during the study period will be assessed using dietary intake data from the average of 3 validated Web-based 24-hour recalls (R24W)
Change in physical activity | 0 to 11 months
  Physical activity during the study period will be assessed primarily using the EPIC-Norfolk Work and leisure time physical activity questionnaire, which categorizes participants into one of 4 groups based on physical activity at work and during leisure time: 1- Inactive, 2- Moderately inactive, 3- moderately active, 4- Active.
Change in sleep quality | 0 to 11 months
  Sleep quality during the study period will be assessed using the Pittsburgh Sleep Quality Index (PSQI) questionnaire with a score varying between 0 and 21; lower score indicates a better sleep quality.
Change in health-related quality of life | 0 to 11 months
  Quality of life during the study period will be assessed using the Short form (SF)-36 health-related quality of life questionnaire, which yields eight subscale scores that are analyzed individually: physical function, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health. Each subscale has a score varying between 0 and 100; higher scores indicate a better quality of life for each individual subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, Principal Investigator — University Laval
Locations (1):
- Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No